CLINICAL TRIAL: NCT00127088
Title: A Prospective Phase II of Peri-Operative Docetaxel + Laparoscopic Radical Prostatectomy in Patients With Localized Gleason 7 pT2a-pT2b Adenocarcinoma and a Risk of Relapse After Radical Prostatectomy
Brief Title: Study of Peri-Operative Docetaxel Plus Laparoscopic Radical Prostatectomy in Prostate Cancer Patients
Status: Suspended | Phase: Phase 2 | Type: Interventional
Sponsor: Gustave Roussy, Cancer Campus, Grand Paris (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Peri-op
Record Dates: First submitted 2005-08-03; First posted 2005-08-05 (Estimated); Last update posted 2006-09-11 (Estimated); Status verified 2006-09

CONDITIONS: Prostate Cancer
Keywords: Patients with localized Gleason 7 pT2a-pT2b adenocarcinoma of the prostate
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Docetaxel

INTERVENTIONS:
Drug: docetaxel
Procedure: laparoscopic radical prostatectomy

SUMMARY:
This is a prospective phase II study of peri-operative docetaxel plus laparoscopic radical prostatectomy in patients with localized Gleason 7 pT2a-pT2b adenocarcinoma of the prostate and a risk of relapse after radical prostatectomy.

ELIGIBILITY:
Inclusion Criteria:

* Patients older than 18 years and less than 70 years
* Histologically-proven Gleason 7 adenocarcinoma of the prostate
* pT2a or pT2b disease based on biopsies of the prostate
* More than 2/3 of positive biopsies or 15 ≤ serum PSA <20
* No previous carcinoma, except basal-cell carcinoma of the skin
* Adequate renal function: measured or calculated creatinine clearance> 60 ml/min
* Absolute granulocyte count ≥ 1,500/mm3, platelets ≥ 100,000 mm3, bilirubin ≤ 1.5 fold the upper normal value
* Signed informed consent.

Exclusion Criteria:

* Patients infected by the Human Immunodeficiency Virus (HIV)
* Contra-indication to general anesthesia or surgery
* Patients who do not fit inclusion criteria

Ages: 18 Years to 70 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37
Dates: Start 2004-10

PRIMARY OUTCOMES:
Complete prostate specific antigen (PSA) response rate

SECONDARY OUTCOMES:
Toxicity
Pathological response rate
Progression free survival
Overall survival

CONTACTS AND LOCATIONS:
Overall Officials: Karim Fizazi, Dr, Principal Investigator — Gustave Roussy, Cancer Campus, Grand Paris
Locations (1):
- Institut Gustave Roussy, Villejuif, France